CLINICAL TRIAL: NCT05079061
Title: A Randomized Controlled Trial of Sublingual Misoprostol in Addition to Routine Uterotonics to Reduce Primary Postpartum Haemorrhage in Low Risk Women After Vaginal Delivery
Brief Title: A Trial of Sublingual Misoprostol to Reduce Primary Postpartum Haemorrhage After Vaginal Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Diana Man-Ka Chan, Associate consultant, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UW 20-044
Record Dates: First submitted 2021-07-01; First posted 2021-10-15 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Primary Postpartum Hemorrhage; Misoprostol; Delivery Complication
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol group (Active Comparator): At delivery of baby, routine uterotonics (syntometrine 1ml intramuscular or syntocinon 5 units intravenous bolus followed by 40 units in 500ml normal saline infusion over 4 hours in women contraindicated for syntometrine) will be given as routine practice, and sublingual misoprostol will be given to women in misoprostol group.
  Interventions: Drug: Misoprostol
- Control group (No Intervention): At delivery of baby, routine uterotonics (syntometrine 1ml intramuscular or syntocinon 5 units intravenous bolus followed by 40 units in 500ml normal saline infusion over 4 hours in women contraindicated for syntometrine) will be given as routine practice, and no additional sublingual misoprostol will be given to women in control group.

INTERVENTIONS:
Drug: Misoprostol — sublingual misoprostol 600 micrograms in addition routine uterotonics at third stage of labour
  Other Names: cytotec
  Arms: Misoprostol group

SUMMARY:
The objective of the randomized controlled study is to compare combination of sublingual misoprostol and routine uterotonics versus routine uterotonics alone on PPH in low risk women after vaginal delivery. The hypothesis is that combination of sublingual misoprostol and routine uterotonics is more effective than routine uterotonics alone in reduction of PPH in low risk women after vaginal delivery.

DETAILED DESCRIPTION:
The investigators propose a multi-center randomized controlled trial. All women eligible for the trial will be recruited at antenatal clinic or antenatal ward. Women with risk factors for PPH and who are planning for Caesarean delivery will be excluded. Women are informed of the study in the antenatal clinic between 36 to 40 weeks gestation. An information sheet will be distributed and a written consent will be obtained. This trial will involve three maternity units in Hospital Authority (Queen Mary Hospital, Queen Elizabeth Hospital and Pamela Youde Nethersole Eastern Hospital) with total annual delivery of 11673 in 2018. Among the annual delivery of 11000, 70% would be vaginal delivery and 60% of women with vaginal delivery would be at low risk for PPH, about 4600 women per year will be eligible in the three units. The investigators aim to recruit 400-500 women per year in total in the three units and the sample size is 1300 women in total over three years.

Eligible women will be randomly assigned in a 1:1 ratio by a computer-generated list to misoprostol or control group when the women are in active labour. Women in misoprostol group will receive sublingual misoprostol 600 micrograms in addition to routine uterotonics, whereas women in control group will receive routine uterotonics. Central randomization will be performed, generated by stratified block randomization, stratified by individual centers. Randomization will be performed when women are in advanced labour i.e. cervical dilatation at 8cm or more and will be stratified by centres and parity (nulliparous vs multiparous).

Antenatal and intrapartum care of the women will follow routine care. A blood sample for complete blood count will be taken when women are admitted in labour. Active management of third stage of labour will be provided as routine postpartum care (including use of routine uterotonics and controlled cord traction). Delayed cord clamping is allowed at discretion of managing clinicians. Studies have shown the delayed cord clamping is beneficial to newborn and it does not increase risk of maternal bleeding. At delivery of baby, routine uterotonics (syntometrine 1ml intramuscular or syntocinon 5 units intravenous bolus followed by 40 units in 500ml normal saline infusion over 4 hours in women contraindicated for syntometrine) will be given as routine practice, and sublingual misoprostol will be given to women in misoprostol group.

Blood loss will be measured during vaginal delivery by direct collection of blood with a calibrated obstetric drape. The calibrated under-buttock drape folds out into a 1x1 meter sterile surface for delivery. The device allows for blood to be collected into a transparent calibrated pouch with capacity up to 2500ml. There are markings on the pouch that aid blood volume measurement. Immediately after delivery of baby and before delivery of placenta, amniotic fluid will be drained and a surgical drape with a graduated bag will be placed under women's buttock to collect the blood loss. The bag will remain in place for at least 15 minutes and until the birth attendants consider that the bleeding has stopped. Swabs and drapes soaked with blood will be weighed using a standardized scale for blood loss calculation (subtracting the known dry weight of the drapes and swabs) in addition to that collected in the graduated bag. Clinicians who assess the blood loss will be blinded to study group allocation. Maternal blood pressure, pulse and temperature will be recorded every 4 hours for one day after delivery. An observation form will be used to record maternal side effects. Blood will be checked for complete blood count on day 2 after delivery.

In order to standardize various study procedures, training will be provided at individual study sites by investigators. Training will include recruitment procedure, randomization , administration of study drug and blood loss measurement method. Research assistant will have regular visit in various study sites to check consistency of the above procedures.

Investigators will have regular communication and meetings with co-investigators at the study sites to review study procedures and to review study progress and address potential problems arising from the study.

ELIGIBILITY:
Inclusion Criteria:

* All women age ≥ 18 years (age of legal consent)
* Singleton pregnancy >= 34 weeks

Exclusion Criteria:

* Women planning for Caesarean section
* Women with known risk factors for PPH, including grand multiparity (>=4), multiple pregnancy, fibroid with size >4cm, history of PPH, placenta previa, large-for-gestational age fetus (defined as EFW >90th centile), polyhydramnios, and previous Caesarean section.
* Women with bleeding tendency or thrombocytopenia < 100 x 109/L
* Women on anticoagulant or aspirin
* Women in whom use of misoprostol / syntocinon / syntometrine is contraindicated
* Women with known hypersensitivity to misoprostol / syntocinon / syntometrine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of primary postpartum haemorrhage | within first 24 hours after delivery
  blood loss 500ml or more at delivery

SECONDARY OUTCOMES:
Percentage of severe postpartum haemorrhage | within first 24 hours after delivery
  blood loss 1000ml or more
Percentage of need for additional uterotonics for treatment of postpartum haemorrhage | within first 24 hours after delivery
  including additional use of syntometrine, syntocinon, carboprost and misoprostol
Duration of third stage of labour | within first 24 hours after delivery
  Time interval between delivery of baby and delivery of placenta
Percentage of need for manual removal of placenta | within first 24 hours after delivery
  Need for manual removal of placenta due to retained placenta
Incidence of uterine atony | within first 24 hours after delivery
  incidence of uterine atony
Change in haemoglobin level (g/dL) after delivery | within 7 days after delivery
  compared with pre-delivery haemoglobin
Change in haematocrit level (L/L) after delivery | within 7 days after delivery
  compared with pre-delivery haematocrit level
Percentage for need for blood transfusion | within 7 days after delivery
  need for blood transfusion due to primary postpartum haemorrhage
Duration of hospital stay after delivery | upto 6 weeks postpartum
  Number of days of hospital stay after delivery due to primary postpartum haemorrhage
Number of participants with side effects | within 7 days after delivery
  Including nausea, vomiting, diarrhea, headache, abdominal pain, metallic taste, high blood pressure (defined by persistently high blood pressure >=140/90mmHg), shivering, pyrexia (>38.5C)
Percentage of maternal infection | within 7 days after delivery
  Positive microbiological cultures in high vaginal swab / endocervical swab / blood culture or clinical infection treated by a course of antibiotics
Patient satisfaction | within 7 days of delivery
  Patient satisfaction regarding the use of sublingual misoprostol by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Diana Man Ka Chan, MBBS, Principal Investigator — Department of Obstetrics & Gynaecology, Queen Mary Hospital

IPD SHARING:
Plan to Share IPD: No